CLINICAL TRIAL: NCT01229072
Title: Clinical Study to Assess the Safety of the Use of the Drug Heparin Sodium Produced by the Laboratory Blausiegel Compared in Parallel to the Product Liquemine ® Laboratory Roche in Patients With Chronic Renal Failure.
Brief Title: Safe Use of Heparin Sodium in Patients With Chronic Renal Failure.
Acronym: Heparin
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Principal Investigator, Azidus Brasil, Principal Investigator Dr. Alexandre Frederico, Azidus Brasil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEPBLA0108
Record Dates: First submitted 2008-10-01; First posted 2010-10-27 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Chronic Renal Failure
Keywords: Safety; Non-inferiority
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Heparin Blausiegel
  Interventions: Biological: Heparin sodic
- 2 (Active Comparator): Liquemine
  Interventions: Biological: heparin liquemine

INTERVENTIONS:
Biological: Heparin sodic — Heparin sodic 150UI/kg
  Arms: 1
Biological: heparin liquemine — Heparin sodic 150UI/kg
  Arms: 2

SUMMARY:
The Heparin form a complex with a plasma protein, antithrombin III (ATIII), which is an endogenous anticoagulant. This complex inhibits the formation of thrombin and accelerates its destruction. Moreover, heparin and other proteases ATIII inactivate the clotting cascade, especially the anti-activated factor X. The end result of these actions is the inhibition of biochemical training and synthesis of certain clotting factors that activators of critical functions in the genesis of a blood clot. Patients with chronic renal failure (CRF) who use the treatment of hemodialysis need a system of anticoagulation with the direct thrombin inhibitor and / or heparinóides to prevent thrombosis.

Based on clinical studies, to control the level of plasma heparin in patients with CRF is essential. Evidence of clotting as APTT, TP, ACT and proof of the activity of anti-factor Xa should be used as a substrate of protection for those patients on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, regardless of color or social class;
* Age above 18 years;
* Patients who agree to participate in the study and signed the free and informed consent (attached);
* Insufficient patients in chronic renal dialysis scheme (3 times per week);
* Low Chronic Renal indication of anticoagulant during dialysis.

Exclusion Criteria:

* Not agree to the terms described in informed consent;
* Patients with sensitivity to heparin sodium;
* Volunteer search with hypersensitivity to benzyl alcohol;
* Patients with a history of bleeding or change in blood clotting that can aggravate or terminate the clinical picture, such as tables of gastric ulcer;
* Patients with a history of peptic ulcer;
* Patients with cancer of any etiology, because of the possibility of compromising the function of the variable coagulation;
* Patients in a period of pregnancy and postpartum;
* Individuals with genetic abnormality of clotting system;
* Patients polytraumatized;
* Patients in use of glucocorticoids for at least 1 month;
* Patients in use of other anticoagulants;
* Patients with high rate of bleeding;
* Patients undergo any surgery performed less than 15 days because of the risk of the formation of hematomas at the site of surgery;
* Patients in use of drugs that affect the hemostasis;
* In addition to these, clinical characteristics that the medical criteria, can interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07

PRIMARY OUTCOMES:
Safety use of the heparin in patients with renal failure. | 12 dialysis sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil